CLINICAL TRIAL: NCT02254590
Title: Irrigation Endoscopic Decompressive Laminotomy. A New Endoscopic Approach for Spinal Stenosis Decompression
Brief Title: Irrigation Endoscopic Decompression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, hesham magdi soliman, Lecturer of Orthopedic Surgery, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Kasr Einy
Record Dates: First submitted 2014-09-26; First posted 2014-10-02 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-09

CONDITIONS: Lumbar Spinal Canal Stenosis
Keywords: IEDL; irrigation endoscopic decompressive laminotomy; irrigation endoscopic decompression; minimally invasive spine surgery; endoscopic decompression; spinal stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IEDL (Experimental): Endoscopic decompression of spinal stenosis
  Interventions: Procedure: Irrigation Endoscopic Decompressive Laminotomy

INTERVENTIONS:
Procedure: Irrigation Endoscopic Decompressive Laminotomy — 2 portals 0.5cm were used one for the endoscope and the other for instruments. For every additional level one portal is added. The endoscope and instruments are directly placed over the surface of lamina without any dissection and saline under pump pressure is used to open a potential working space. Unilateral laminotomy/laminectomy is performed according to the severity of stenosis, followed by bilateral decompression beneath the midline structures.

SUMMARY:
To evaluate a new endoscopic technique for lumbar spinal canal decompression.

DETAILED DESCRIPTION:
104 consecutive patients suffering of neurogenic claudication were included in the study.

Patients were operated using the irrigation endoscopic decompression technique. Mean Follow up was 28 months Primary outcome measures were assessed using the Oswestry Disability Index [19] and the modified Macnab Criteria All statistical calculations were done using computer programs SPSS (Statistical Package for the Social Science; SPSS Inc., Chicago, IL, USA) version 15 for Microsoft Windows

ELIGIBILITY:
Inclusion Criteria:

1. Neurogenic claudication or radicular leg pain with or without back pain, and/or a neurological deficit
2. Symptoms and signs correlating with moderate to severe spinal canal stenosis as shown on MRI. (Degenerative and congenital bony stenosis were included)
3. Failure of 3 months conservative treatment
4. Grade I degenerative spondylolisthesis and degenerative scoliosis

Exclusion Criteria:

1. Segmental Instability
2. Lytic Spondylolisthesis

2- Predominant low back pain

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2009-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index | 24 months
  Measurement of pain intensity, personal care, sitting, standing, walking, lifting,sleeping, sex life, social life, travelling
Modified Macnab criteria | 24 months
  patient satisfaction, the need for medications, ability to return to activity

SECONDARY OUTCOMES:
Time for ambulation | 72 hours
  postoperative time required to start ambulation
Time for hospitalization | 72 hours
  postoperative hospital stay till discharge
VAS for back pain | 72 hours
  Pain intensity on scale from 0-10